CLINICAL TRIAL: NCT04031521
Title: Near-infrared Spectroscopy in Sickle Cell Pediatric Patients During Pain Crisis and After Recovery
Brief Title: Near Infrared Spectroscopy in Sickle Cell Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patient were available/ found
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Suvankar Majumdar, Chief of Hematology, Children's National Research Institute
Other Study IDs: Pro00012424
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Sickle cell pain crisis
  Interventions: Diagnostic Test: Near infrared spectroscopy
- Sickle cell steady-state
  Interventions: Diagnostic Test: Near infrared spectroscopy

INTERVENTIONS:
Diagnostic Test: Near infrared spectroscopy — NIRS is an emerging technology for measuring tissue oxygenation and endothelial function. NIRS light can penetrate through biological tissues, including skin, bone, and muscle. Similar to other optical methods, light is applied to the region of interest and undergoes scattering and absorption before being detected by a photosensor. This technique is commonly used to assess oxygen availability and consumption in living tissues. Using different wavelengths, NIRS can differentiate between oxygenated and deoxygenated hemoglobin in blood and can measure changes in total hemoglobin concentration, using the sum of oxygenated and deoxygenated hemoglobin.

SUMMARY:
Endothelial dysfunction contributes to vaso-occlusion and acute pain in sickle cell disease. Near infrared spectroscopy (NIRS) technology can measure tissue oxygenation and endothelial function. The main objective of this study is to study the natural history of tissue muscle oxygenation using NIRS in pediatric sickle cell subjects experiencing acute pain and pediatric sickle cell patients in steady-state.

ELIGIBILITY:
Inclusion Criteria for Subjects with Sickle Cell Disease in Pain Crisis:

1. Age 6 to 21 years old.
2. Diagnosis of sickle cell anemia: a. Diagnosis of sickle cell disease (electrophoresis or HPLC documentation of hemoglobin SS, SC, S-beta-thalassemia or other hemoglobinopathies causing sickle cell disease is required).
3. Acute onset pain crisis in a distribution typical for that subject, onset within the last 7 days and for which hospitalization and parenteral narcotic pain treatment are required.
4. Ability to provide informed written consent.

Exclusion Criteria for Subjects with Sickle Cell Disease in Pain Crisis:

1. Pregnancy.
2. History of non-trivial injury, burns, surgery or skin ulcers on the arms.
3. Fever or suspected sepsis at time of pain crisis
4. Administration of any of the following drugs within the last 14 days:

   * Phosphodiesterase-5 inhibitors (sildenafil, vardenafil, tadalafil)
   * Endothelin-1 receptor blockers (bosentan, sitaxentan, ambrisentan, tezosentan)
   * Nitric oxide donors (nitroglycerin, nitroprusside, nitrates)
5. Ingestion of caffeine within the 12 hours before the start of the study appointment, or tobacco use within the 30 days before the study appointment.
6. Diagnosis with any of the following chronic diseases or conditions:

   * History of high blood pressure
   * History of high cholesterol
   * History of diabetes
   * History of chronic kidney disease (serum creatinine must not be greater than 2 mg/dL)
   * History of coronary artery disease or peripheral vascular disease
7. Received a blood transfusion within 7 days of the study procedure.

Inclusion Criteria for Subjects with Sickle Cell Disease in Steady State:

1. Age 6-21 years
2. Diagnosis of sickle cell disease (electrophoresis or HPLC documentation of hemoglobin SS, SC, S-beta-thalassemia or other hemoglobinopathies causing sickle cell disease is required).
3. Ability to provide informed written consent.

Exclusion Criteria for Subjects with Sickle Cell Disease in Steady State:

1. Pregnancy.
2. History of non-trivial trauma, burns, surgery or skin ulcers on the arms.
3. Fever or suspected sepsis at time of pain crisis
4. Experience of an acute pain crisis requiring intravenous (IV) narcotics and hospital admission within the last 14 days.
5. Ingestion of caffeine within the 12 hours before the start of the study appointment, or tobacco use within the 30 days before the study appointment.
6. Administration of any of the following drugs within the last 14 days:

   * Phosphodiesterase-5 inhibitors (sildenafil, vardenafil, tadalafil)
   * Endothelin-1 receptor blockers (bosentan, sitaxentan, ambrisentan, tezosentan)
   * Nitric oxide donors (nitroglycerin, nitroprusside, nitrates)
7. Diagnosis of any of the following chronic diseases or conditions:

   * History of high blood pressure
   * History of high cholesterol
   * History of diabetes
   * History of chronic kidney disease (serum creatinine must not be greater than 2 mg/dL)
   * History of coronary artery disease or peripheral vascular disease
8. Received a blood transfusion within 7 days of the study procedure.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects 6 to 21 years of age of all sickle cell genotypes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation | 6 months

SECONDARY OUTCOMES:
Nitric oxide | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No